CLINICAL TRIAL: NCT01027156
Title: The Influence of a High Intensity Physical Activity Intervention on a Selection of Health Related Outcomes: An Ecological Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of Scotland (Other)
Collaborators: Swansea University (Other)
Responsible Party: Duncan Buchan, Lecturer, University of the West of Scotland
Purpose: Prevention
Other Study IDs: HI Intervention
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: To Assess the Impact of the HIT Intervention on Physiological Responses; To Assess the Role of a Secondary High School as a Setting for Promoting Healthy Eating and PA Behaviours; To Determine the Associations Between CVD Risk Factors at Baseline in 15 - 18 Year Old Youth
Keywords: Public Health; Biochemistry; Ecological
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Intensity Exercise (Experimental)
  Interventions: Behavioral: High Intensity Exercise

INTERVENTIONS:
Behavioral: High Intensity Exercise — In this study, participants will be instructed to sprint maximally for a period of 30 seconds. Following 30s rest, the participants will be instructed to repeat this procedure a further 3 times. This equates to 2 minutes of maximal effort sprinting interspersed with 2 minutes recovery. Participants will be requested to perform this protocol 3 times weekly. Training progression will be implemented by increasing the number of repeats from four repetitions during weeks 1 and 2, to five repetitions during weeks 3 and 4, to six repetitions during weeks 5 and 6. Finally, during week 7 participants will still perform six repetitions but interspersed by only 20 s recovery.

SUMMARY:
The purpose of this study is to determine whether a High Intensity exercise intervention can elicit cardiovascular disease protection in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 15 - 18 yer old that are capable of performing vigorous exercise

Exclusion Criteria:

* Any health condition that would prevent them from undertaking vigorous exercise

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To improve blood lipid profiles and lower levels of plasma inflammatory markers.

SECONDARY OUTCOMES:
To determine the associations between CVD risk factors at baseline in 15 - 18 year old youth.

CONTACTS AND LOCATIONS:
Locations (1):
- Holy Cross High School, Hamilton, South Lanarkshire, United Kingdom

REFERENCES:
- [Derived] Buchan DS, Ollis S, Young JD, Cooper SM, Shield JP, Baker JS. High intensity interval running enhances measures of physical fitness but not metabolic measures of cardiovascular disease risk in healthy adolescents. BMC Public Health. 2013 May 24;13:498. doi: 10.1186/1471-2458-13-498. PMID 23705968
- [Derived] Buchan DS, Ollis S, Thomas NE, Baker JS. The influence of a high intensity physical activity intervention on a selection of health related outcomes: an ecological approach. BMC Public Health. 2010 Jan 8;10:8. doi: 10.1186/1471-2458-10-8. PMID 20064208